CLINICAL TRIAL: NCT03546452
Title: A Prospective Study to Evaluate the Results of Different NGS- Panels in Mutation Detection and Tumor Mutation Burden(TMB) Calculation by Using Malignant Hydrothorax From NSCLC
Brief Title: A Prospective Study to Evaluate the Consistency of Next-Generation Sequencing(NGS)-Panels by Using Malignant Hydrothorax Form NSCLC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Sinotech Genomics Co., Ltd (Unknown); Amoy Diagnostics (Industry); Guangzhou Burning Rock Medical Examination Institute Co., Ltd. (Industry); Geneplus-Beijing Co. Ltd. (Industry); Berry Genomics Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Lu Shun, Shanghai Chest Hospital, Shanghai Chest Hospital
Other Study IDs: shanghai Chest 0014
Record Dates: First submitted 2018-05-22; First posted 2018-06-06 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Malignant Hydrothorax; NSCLC
Keywords: NSCLC; malignant hydrothorax; prospective study

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cell block obtain from malignant NSCLC hydrothorax
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- malignant NSCLC hydrothorax: cell free DNA ,which is purified from malignant NSCLC hydrothorax, tested by in vitro NGS-panel
  Interventions: Diagnostic Test: in vitro NGS-panel

INTERVENTIONS:
Diagnostic Test: in vitro NGS-panel — cell free DNA ,which was purified from hydrothorax, is used to be tested by NGS-panel

SUMMARY:
A prospective study to evaluate consistency of different NGS-panel. Cell free DNA is purified from each malignant hydrothorax from NSCLC .Different NGS-panels are applied to perform in vitro diagnosis to detect Single Nucleotide Variants(SNV) and to calculate TMB value in these DNA samples.Consistency of enrolled NGS-panels are then evaluated by statistical analysis.

DETAILED DESCRIPTION:
1. Chest Hospital in accordance with the clinical requirements of the treatment required to extract ML hydrothorax sent to hospital pathology department for exfoliated Cell diagnosis and production of cell wax block, while the additional responsibility for the extraction of hydrothorax 500ml, and collect 10ml venous blood sample, Venous blood samples are stored in either the A cell-free DNA Blood collection Tube (STRECK tube) or the ethylenediaminetetraacetic acid(EDTA) anticoagulant tube.
2. Amoy Diagnostics Co., Ltd. (AmoyDx) is responsible for plasma separation after sampling 2 hours, plasma is frozen by the chest Hospital, AmoyDx completes the purification of peripheral blood cells genomic DNA , and which is divided into 6 parts ,5 of which are send to in vitro diagnostic products (IVD) enterprises to perform NGS-Panel detection.
3. 100ml hydrothorax is send to each IVD enterprise.
4. Each IVD enterprise carries on the hydrothorax cell free DNA and peripheral blood cell genomic DNA NGS-Panel detection according to their own protocol.
5. Each IVD enterprise will complete the test within 7-10 working days and fill out the results in accordance with the report template provided by this research project (provided by Guangzhou Burning Rock Medical Examination Institute Co., Ltd.) and submit to sponsor by email.
6. Sponsor would use whole exon panel (WES) to obtain an TMB value if needed.
7. Employ four-grid analysis to evaluate positive compliance rate, negative compliance rate, total compliance rate of all submitted data.
8. Employ kappa test to evaluate the consistency of each two detections.

ELIGIBILITY:
Inclusion Criteria:

* Advanced malignant lung cancer, with treatment of pleural effusion, hydrothorax volume not less than 800ml

Exclusion Criteria:

* The sample size is not sufficient to detect.
* There are not enough tumor cells in the tissue section to be evaluated through the pathology department of the chest Hospital.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients in shanghai chest hospital
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-05-18 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate consistency of TMB value of different NGS-Panel | 5 months
  All DNA samples were tested to calculate TMB value by all enrolled NGS-panel (include WES if necessary), each sample is then to be marked as TMB high, TMB median or TMB low according to the cutoff value identified by different IVD enterprises.
  Employ Cohen's kappa test to calculate the kappa value to measures inter-rater agreement for categorical result.

CONTACTS AND LOCATIONS:
Overall Officials: shun lu, Prof., Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shangha Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided